CLINICAL TRIAL: NCT05088304
Title: The Application Value of Preoperative Fat-free Mass Index Within GLIM-defined Malnutrition Criteria for Postoperative Outcomes in Patients With Esophagogastric Cancer
Brief Title: GLIM-defined Malnutrition Criteria for Postoperative Outcomes in Patients With Esophagogastric Cancer
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Collaborators: Jiangsu Cancer Institute & Hospital (Other); Subei People's Hospital of Jiangsu Province (Other); Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Wang Xinying, Professor, Jinling Hospital, China
Other Study IDs: JinlingHospital-1; 201502022 (Other Grant/Funding Number: Research Special Fund for Public Welfare Industry of Health)
Record Dates: First submitted 2021-09-20; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Cancer of Stomach; Cancer of Esophagus; Malnutrition; Muscle Loss
Keywords: FFIM; GLIM; Cancer; Postoperative complications
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Malnutrition; Muscular Atrophy; Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The normal FFMI group: The FFMI was calculated as follows: FFMI = fat-free mass (kg)/height squared (m2). FFMI cut-off values (derived from BIA measurements, </≥15 kg/m2 for females and </≥17 kg/m2 for males). Patients with esophagogastric cancer were then divided into the normal FFMI group (FFMI ≥17 kg/m2 for male and FFMI ≥15 kg/m2 for female).
  Interventions: Other: no intervention
- The low FFMI group: The FFMI was calculated as follows: FFMI = fat-free mass (kg)/height squared (m2). FFMI cut-off values (derived from BIA measurements, </≥15 kg/m2 for females and </≥17 kg/m2 for males). Patients with esophagogastric cancer were then divided into the low FFMI group (FFMI <17 kg/m2 for male and FFMI <15 kg/m2 for female).
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The present study aims to investigate the prognostic value of preoperative fat-free mass index for postoperative outcomes in patients undergoing esophagogastric cancer surgery, and to explore the role of the FFMI in the Global Leadership Initiative on Malnutrition (GLIM) criteria.

DETAILED DESCRIPTION:
The GLIM criteria of malnutrition as a consensus lack of optimal combination in clinical validation. After the publication of the GLIM consensus, few studies have examined the effect of reduced FFMI on the clinical prognosis of patients with esophagogastric cancer, and whether the FFMI can be used as an effective diagnostic criterion of malnutrition in esophagogastric cancer needs to be further studied.

Therefore, the present study aims were to investigate the prognostic value of preoperative fat-free mass index for postoperative outcomes in patients undergoing esophagogastric cancer surgery, and to explore the role of the FFMI in the GLIM consensus for malnutrition.

ELIGIBILITY:
Inclusion Criteria:

Elective surgery for esophagogastric cancer (there was a clear pathological diagnosis before surgery); NRS2002≥3; Preoperative BIA examination was performed.

Exclusion Criteria:

Discharged from a hospital within 24 hours; No BIA examination and not suitable for BIA examination (such as ascites, edema, amputation and pace-maker); Hepatic insufficiency (alanine transaminase/aspartate transaminase ratio 200% above normal range or bilirubin>3mg/dL) ; Renal insufficiency (serum creatinine>1.5mg/dL); Emergency operation; Pregnancy; Missing the postoperative information follow-up data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective surgery for esophagogastric cancer (there was a clear pathological diagnosis before surgery)
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
postoperative complications | Within 60 days after surgery
  postoperative complications (infectious complications and noninfectious complications)

SECONDARY OUTCOMES:
length of stay (LOS) | Within 60 days after surgery
  length of stay (LOS)
wound healing time | Within 60 days after surgery
  wound healing time
postoperative antibiotic time | Within 60 days after surgery
  postoperative antibiotic time
nutritional status | up to 4 weeks
  nutritional status ( such as: weight，albumin，prealbumin)
hospitalization cost | Within 60 days after surgery
  hospitalization cost(including: surgery and medicine costs)